CLINICAL TRIAL: NCT01540123
Title: The Time Effects of a Berry Extract Upon Cerebral Blood Flow.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: The New Zealand Institute of Plant and Food Research Ltd. (Other Government)
Responsible Party: Principal Investigator, Anthony Watson, Principal Investigator, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 28AI3
Record Dates: First submitted 2012-02-06; First posted 2012-02-28 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Cerebral Blood Flow

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Sugar matched control containing no phytochemicals
  Interventions: Dietary Supplement: Control
- Berry drink standardised to contain 500mg of polyphenols (Experimental): Cold pressed berry drink standardised to contain 500mg of berry polyphenols
  Interventions: Dietary Supplement: Berry drink

INTERVENTIONS:
Dietary Supplement: Berry drink — Cold pressed berry drink standardised to contain 500mg of berry polyphenols
  Arms: Berry drink standardised to contain 500mg of polyphenols
Dietary Supplement: Control — Sugar matched control containing berry flavouring and no phytochemicals
  Arms: Control

SUMMARY:
Berry fruits are widely recognised as natural functional food products. They contain several different phytochemicals which have potential to modulate human health and wellbeing. There is however some debate regarding the mechanisms driving their health promoting properties.

Despite the wide health promoting properties of fruit extracts reported in the literature, considerable interest over the past decade has primarily been focused on their roles in reducing risk factors associated with cancer and heart disease. Consequently, there remains a paucity of actual scientific information on their role in modulating brain functions, such as mood, learning and memory, any decrements of which have very negative impacts on the quality of life.

Fruit phytochemicals from other sources have been shown to mediate both peripheral and cerebral blood flow. However, a modulation of cerebral blood flow has not been shown with berries as yet. Cerebral blood flow must be maintained to ensure a constant delivery of oxygen and glucose as well as the removal of waste products. The modulation of cerebral blood flow via supplementation of berry polyphenols could therefore be a potential way to positively modulate human cognitive behavior. The link between acute increases in cerebral blood flow and increased cognition is currently a little weak but it could give a good platform for long term behavioral and health benefits via increased cerebral/peripheral blood flow and decreased MAO-B activity.

The aims of the study are therefore to investigate the impact of the berry extract on digital volume pulse, blood pressure and cerebral blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* none smokers
* aged between 18 and 35 years

Exclusion Criteria:

* History of neurological, vascular or psychiatric illness.
* Current diagnosis of depression and/or anxiety.
* History or current diagnosis of drug/alcohol abuse.
* Anaemia.
* Any heart disorder.
* Hypertension
* Any respiratory disorder.
* Diabetes.
* Food intolerances/sensitivities.
* Phenylketonuria.
* Use tobacco products or have ceased in the last 6 months.
* Currently taking any prescribed, illicit or herbal drugs.
* Any known active infections.
* HIV antibody positive.
* Currently have, have ever had, or may be at risk of hepatitis.
* Have suffered from jaundice within the last year.
* Have haemophilia or any similar clotting disorder.
* History of head trauma
* History of migraines
* History of learning difficulties
* Any Issues with giving blood samples.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Digital Volume Pulse | Change from baseline at 15, 30, 45, 60, 100, 120, 150, 180, 240 minutes and 24 hours post dose
Cerebral blood flow | Continuous measure from baseline to 100 minutes post dose
Blood platelet MAO-B activity | Change from baseline at 15, 30, 45, 60, 100, 120, 150, 180, 240 minutes and 24 hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Brain, Performance and Nutrition Research Centre, Newcastle upon Tyne, Newcastle Upon-Tyne, United Kingdom

REFERENCES:
- [Derived] Watson AW, Scheepens A, Kennedy DO, Haskell-Ramsay CF. Effects of blackcurrant juice on pre-frontal cortical haemodynamics and cognition in healthy young adults. Nutr Neurosci. 2026 Jan;29(1):14-28. doi: 10.1080/1028415X.2025.2538062. Epub 2025 Sep 25. PMID 40999681
- See also: Related Info — http://www.nutrition-neuroscience.co.uk/